CLINICAL TRIAL: NCT06272695
Title: Glucagon Rescue of Insulin-Induced Hypoglycemia in Adults With Type 1 Diabetes Treated With Volagidemab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: REMD Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R477-203
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — volagidemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 35 mg Volagidemab (Experimental): Volagidemab 35 mg will be administered by subcutaneous (SC) injection once weekly for 6 weeks.
  Interventions: Biological: Volagidemab

INTERVENTIONS:
Biological: Volagidemab — Administered by SC injection once weekly for 6 weeks

SUMMARY:
This trial is designed to evaluate the effect of glucagon receptor antagonism by volagidemab (once weekly) on glucose recovery from hypoglycemia after treatment with glucagon in adults with type 1 diabetes. After informed consent, Screening procedures to establish subject eligibility will be performed within a period of 28 days. Approximately 24 subjects with type 1 diabetes mellitus (T1DM) on stable doses of insulin will be enrolled.

After enrollment, subjects will undergo a baseline Hypoglycemia Recovery Procedure (with glucagon rescue). Subjects will then receive volagidemab subcutaneously (SC) once weekly for 6 weeks. At the end of the treatment phase, subjects will undergo a second Hypoglycemia Recovery Procedure. Subjects will be followed for 6 weeks after the last volagidemab dose with a final End-of-Study (EOS) visit during Week 12. The primary outcome will be the change in time to glucagon treatment success at Week 6 versus baseline.

ELIGIBILITY:
Inclusion Criteria:

* Receiving insulin for the treatment of documented diagnosis of T1DM for at least 2 years
* Body Mass Index (BMI) of 18.5 kg/m2 to 35.0 kg/m2
* On treatment with a stable insulin regimen for at least 8 weeks
* Currently using a continuous glucose monitoring (CGM) system
* HbA1c less than or equal to 10.0%
* Females of non-childbearing potential must be ≥1 year post-menopausal or documented as being surgically sterile. Females of childbearing potential must agree to use two methods of contraception during the entire study and for an additional 3 months after the end of dosing with the investigational product
* Male subjects must be willing to use clinically acceptable method of contraception during the entire study and for an additional 3 months after the end of the treatment period
* Other inclusion criteria may apply.

Exclusion Criteria:

* History of type 2 diabetes, maturity onset diabetes of the young (MODY), pancreatic surgery or chronic pancreatitis
* Pancreas, pancreatic islet cells, or renal transplant recipient
* T1DM treatment with any other antihyperglycemic drug (e.g., metformin, alpha- glucosidase inhibitors, SGLT-2 inhibitors, pramlintide, inhaled insulin, pre-mixed insulins, etc.) within 30 days of Day 1
* Occurrence of severe hypoglycemia involving coma and/or seizure that required hospitalization or hypoglycemia-related treatment by an emergency physician or paramedic within 3 months prior to Day 1
* Myocardial infarction, unstable angina, revascularization procedure, or cerebrovascular accident ≤12 weeks
* Indication of liver disease
* Current signs and symptoms of anemia
* Untreated eating disorders such as bulimia or anorexia nervosa
* History of pancreatitis, pancreatic neuroendocrine tumors or multiple endocrine neoplasia (MEN) or family history of MEN.
* Treatment with systemic corticosteroids within 30 days of Day 1, or planned initiation of such therapy during the study.
* Medical history of cancer or treatment for cancer in the last five years
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Other exclusion criteria may apply

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Time to glucagon treatment success at Week 6. | 6 weeks
  The primary outcome of the study is the change in time to glucagon treatment success, defined as an increase in plasma glucose of ≥20 mg/dL from the glucose nadir after receiving glucagon during insulin-induced hypoglycemia, from baseline to Week 6.

SECONDARY OUTCOMES:
Blood glucose response to glucagon rescue treatment during insulin-induced hypoglycemia. | 6 weeks
  Percentage of subjects achieving glucagon treatment success, defined as an increase in plasma glucose to ≥70 mg/dL or an increase of ≥20 mg/dL from the glucose nadir within 30 minutes of receiving glucagon during insulin-induced hypoglycemia, at Week 6.
Treatment emergent adverse events (AEs) | 12 weeks
  The subject incidence rates of AEs will be tabulated by system organ class, preferred term, and severity grade for all treatment emergent, serious, treatment related, and serious treatment related AEs.
Hypoglycemia symptoms - Edinburgh Hypoglycemia Scale | 6 weeks
  Results of the Edinburgh Hypoglycemia Scale will be summarized over Intent-to-Treat (ITT) set using descriptive statistics by visit (baseline, week 6) and timepoint (baseline, t = 15, 30, 45, and 60 min after glucagon administration for Edinburgh Hypoglycemia Scale). Changes from baseline in Edinburgh hypoglycemia scale will be summarized similarly.
Hypoglycemia symptoms - Clarke Survey | 6 weeks
  Results of the Clarke Survey will be summarized over Intent-to-Treat (ITT) set using descriptive statistics by visit (baseline, week 6). Changes from baseline in Clarke Survey will be summarized similarly.
Hypoglycemia symptoms - Gold Questionnaire | 6 weeks
  Results of the Gold Questionnaire will be summarized over Intent-to-Treat (ITT) set using descriptive statistics by visit (baseline, week 6). Changes from baseline in Gold Questionnaire will be summarized similarly.
Change from baseline in hemoglobin A1c (HbA1c) at Week 6. | 6 weeks
  Change from baseline in hemoglobin A1c (HbA1c) at Week 6, after repeated doses of volagidemab

CONTACTS AND LOCATIONS:
Overall Officials: Zung Thai, MD, Study Director — REMD Biotherapeutics
Locations (2):
- United States (2):
  - Altman Clinical and Translational Research Institute, San Deigo, California
  - Diablo Clinical Research, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: Undecided